CLINICAL TRIAL: NCT00382109
Title: A Randomized Trial of Sirolimus-Based Graft Versus Host Disease Prophylaxis After Hematopoietic Stem Cell Transplantation in Relapsed Acute Lymphoblastic Leukemia
Brief Title: Tacrolimus and Methotrexate With or Without Sirolimus in Preventing Graft-Versus-Host Disease in Young Patients Undergoing Donor Stem Cell Transplant for Acute Lymphoblastic Leukemia in Complete Remission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASCT0431; NCI-2009-01068 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000500131 (Other: Clinical Trials.gov); COG-PBMTC-ONCO51 (Other: Children's Oncology Group); COG-ASCT0431 (Other: Children's Oncology Group); U10CA098543 (NIH)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Results first posted 2017-02-09 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2019-06

CONDITIONS: B-cell Childhood Acute Lymphoblastic Leukemia; Childhood Acute Lymphoblastic Leukemia in Remission; Graft Versus Host Disease; L1 Childhood Acute Lymphoblastic Leukemia; L2 Childhood Acute Lymphoblastic Leukemia; T-cell Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Graft vs Host Disease; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Thiotepa; Cyclophosphamide; Tacrolimus; Methotrexate; merphos; Sirolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacro-MTX/Sirolimus GVHD Prophylaxis Regimen (Experimental): Preparative regimen of total body irradiation (TBI) 200 cGy BID days -8,-7, & -6, Thiotepa IV (dose 5 mg/kg/day on days -5 & -4) & cyclophosphamide IV (dose 60 mg/kg/day on days -3 & -2). Tacrolimus IV (dose 0.02 mg/kg/day) continuously or orally daily on day -2 with a taper starting on day 42 - day 98 (patients undergoing matched sibling donor transplantation) OR tacrolimus IV (dose 0.02 mg/kg/day) continuously or orally daily beginning on day -2 followed by a taper on day 100 through day 180 (patients undergoing other related, unrelated, or cord blood donor transplantation) in the absence of GVHD. Patients also receive methotrexate IV (5 mg/m2/dose) on days 1,3, & 6 (patients with matched sibling and umbilical cord blood donors) OR days 1,3 6, & 11 (patients with other related/unrelated bone marrow and peripheral blood stem cell donors) and oral sirolimus (dose 2.5mg/m2/day - 4 mg max starting dose) daily starting on day 0 followed by a taper starting on day 180 through day 207.
  Interventions: Drug: thiotepa; Drug: cyclophosphamide; Drug: tacrolimus; Drug: methotrexate; Drug: sirolimus; Radiation: total body irradiation
- Tacro-MTX GVHD Prophylaxis (Active Comparator): Preparative regimen of total body irradiation (TBI) 200 cGy BID days -8,-7, & -6, Thiotepa IV (dose 5 mg/kg/day on days -5 & -4) & cyclophosphamide IV (dose 60 mg/kg/day on days -3 & -2). Tacrolimus IV (dose 0.02 mg/kg/day) continuously or orally (when able) daily on day -2 with a taper starting on day 42 - day 98 (patients undergoing matched sibling donor transplantation) OR tacrolimus IV (dose 0.02 mg/kg/day) continuously or orally daily beginning on day -2 followed by a taper on day 100 through day 180 (patients undergoing other related, unrelated, or cord blood donor transplantation) in the absence of GVHD. Patients also receive methotrexate IV (5 mg/m2/dose) on days 1,3, & 6 (patients with matched sibling and umbilical cord blood donors) OR days 1,3 6, & 11 (patients with other related/unrelated bone marrow and peripheral blood stem cell donors).
  Interventions: Drug: thiotepa; Drug: cyclophosphamide; Drug: tacrolimus; Drug: methotrexate; Radiation: total body irradiation

INTERVENTIONS:
Drug: thiotepa — Given IV
  Other Names: Oncotiotepa; STEPA; TESPA; Tespamin; TSPA
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: tacrolimus — Given IV or orally
  Other Names: FK 506; Prograf
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: sirolimus — Given orally
  Other Names: AY 22989; Rapamune; rapamycin; SLM
  Arms: Tacro-MTX/Sirolimus GVHD Prophylaxis Regimen
Radiation: total body irradiation — Part of the transplant preparatory regimen
  Other Names: TBI

SUMMARY:
This randomized phase III trial is studying tacrolimus, methotrexate, and sirolimus to see how well they work compared to tacrolimus and methotrexate in preventing graft-versus-host disease in young patients who are undergoing donor stem cell transplant for intermediate-risk or high-risk acute lymphoblastic leukemia in second complete remission and high risk acute lymphoblastic leukemia in first remission. Giving chemotherapy, such as thiotepa and cyclophosphamide, and total-body irradiation before a donor stem cell transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus, methotrexate, and sirolimus after the transplant may stop this from happening. It is not yet known whether tacrolimus and methotrexate are more effective with or without sirolimus in preventing graft-versus-host disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the post-transplant 2-year event-free survival of pediatric patients with intermediate-risk or high-risk acute lymphoblastic leukemia (ALL) in second complete remission or high risk ALL in first remission undergoing allogeneic hematopoietic stem cell transplantation treated with graft-versus-host disease (GVHD) prophylaxis comprising tacrolimus and methotrexate with or without sirolimus.

SECONDARY OBJECTIVES:

I. Compare rates of relapses, transplant-related mortality, and acute and chronic GVHD in these patients.

II. Evaluate the relative contribution of resistance by ALL blasts to cytolytic therapy (e.g., chemotherapy/irradiation) as a cause of relapse post-transplantation by correlating ALL in vivo blast resistance with in vivo sirolimus, inhibition levels of the mTOR pathway in patients treated with sirolimus, and altered resistance pathways in ALL blasts measured by microarray analysis.

III. Evaluate the relative contribution of resistance by ALL blasts to the donor immune response as a cause of relapse post-transplantation by correlating the development of donor anti-ALL T-cell response, the development of acute and/or chronic GVHD, and the detection of altered ALL blast immunogenicity after transplant with increased minimal residual disease, persistent recipient chimerism, and relapse.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to specific combinations of risk (intermediate CR2 vs high CR2 vs high CR1), donor type (matched sibling vs unrelated or other related), and stem cell source (filgrastim [G-CSF]-primed bone marrow vs unprimed bone marrow vs bone marrow vs peripheral blood vs umbilical cord blood).

PREPARATIVE REGIMEN: Patients undergo total-body irradiation twice daily on days -8 to -6 and receive thiotepa IV on days -5 and -4 and cyclophosphamide IV on days -3 and -2.

ALLOGENEIC HEMATOPOIETIC STEM CELL TRANSPLANTATION: Patients undergo allogeneic hematopoietic stem cell transplantation on day 0.

GRAFT-VERSUS-HOST DISEASE (GVHD) PROPHYLAXIS: Patients are randomized to 1 of 2 treatment arms.

ARM I: (experimental) Patients receive tacrolimus IV continuously or orally (when able) daily beginning on day -2 followed by a taper beginning on day 42 and continuing until day 98 (for patients undergoing matched sibling donor transplantation) OR tacrolimus IV continuously or orally daily beginning on day -2 followed by a taper beginning on day 100 and continuing until day 180 (for patients undergoing related, unrelated, or cord blood donor transplantation) in the absence of GVHD. Patients also receive methotrexate IV on days 1, 3, and 6 (for patients with matched sibling and umbilical cord blood donors) OR days 1, 3, 6, and 11 (for patients with unrelated bone marrow and peripheral blood stem cell donors) and oral sirolimus daily beginning on day 0 followed by a taper beginning on day 180 and continuing until day 207.

ARM II: (control) Patients receive tacrolimus and methotrexate as in arm I.

After completion of study treatment, patients are followed periodically for approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed acute lymphoblastic leukemia (ALL) in second complete remission (CR2) (M1 bone marrow, < 5% blasts by morphology) meeting the following criteria:

  * Intermediate risk relapsed ALL in CR2 (may receive matched sibling transplantation only) meeting 1 of the following criteria:

    * B-lineage ALL in CR2 after a late first bone marrow (BM) relapse (≥ 36 months after the initiation of primary chemotherapy) with or without associated extramedullary disease
    * B-lineage ALL in CR2 after a very early isolated extramedullary relapse (<18 months from the initiation of primary chemotherapy)
  * High risk relapsed ALL in CR2 (may receive other related donor, unrelated donor, or matched sibling transplantation) meeting 1 of the following criteria:

    * In CR2 after an early first BM relapse (< 36 months from initiation of primary chemotherapy)
    * T-lineage ALL in CR2 after a first BM relapse occurring at any time after initiation of primary chemotherapy
    * Philadelphia chromosome-positive ALL in CR2 after a first BM relapse occurring at any time after the initiation of primary chemotherapy
    * T-lineage ALL in CR2 after a very early isolated extramedullary relapse (<18 months from the initiation of primary chemotherapy)
  * High risk de novo ALL in CR1 (may receive matched sibling, other related/unrelated BM/PBSC or unrelated CB transplantation) meeting 1 of the following criteria:

    * Patients with the presence of t(9;22) translocation (Ph+) detected by cytogenetic or PCR analysis at initial diagnosis. For patients on AALL0622, the criteria for transplant are 1) any patient with Ph+ ALL with an available matched sibling donor or 2) any patient with Ph+ ALL that is defined as high risk (MRD > 1% Day 29 or MRD > 0.01% end-Consolidation Block 2) with any available donor, related or unrelated. Patients enrolled on AALL0622 are only eligible if they follow this algorithm.
    * Patients with the presence of extreme hypodiploidy (< 44 chromosomes or DNA index of < 0.81) detected by cytogenetic/ploidy analysis at initial diagnosis.
    * Patients with the presence of 11q23 (MLL) rearrangements detected by cytogenetic or PCR analysis at initial diagnosis who are slow early responders (M2/M3 at Day 14 or MRD > 0.1% at Day 29).
* Enrolled on an appropriate COG relapsed ALL clinical trial after completing the required study therapy (i.e., minimum 1 re-induction course (4-6 weeks) and 1 round of intensive consolidation chemotherapy (3-6 weeks). Patients with high risk ALL in CR1 are eligible as soon as they have achieved a CR.

  * Patients not on a COG relapsed ALL clinical trial are eligible provided they have received ≥ 1 round of re-induction lasting 4-6 weeks and 1 round of intensive consolidation chemotherapy lasting 3-6 weeks
* No B-cell ALL L3 morphology with evidence of myc translocation by molecular or cytogenetic technique
* No Down syndrome
* No evidence of active CNS or other extramedullary disease (i.e., no CNS2)
* Karnofsky performance status (PS) 60-100% (for patients > 16 years of age) OR Lansky PS 60-100% (for patients ≤ 16 years of age)
* Shortening fraction ≥ 27% by echocardiogram OR ejection fraction ≥ 50% by radionuclide angiogram
* ALT or AST < 5 times upper limit of normal
* Bilirubin < 2.5 mg/dL (unless an increase is attributable to Gilbert's syndrome)
* Creatinine clearance OR radioisotope glomerular filtration rate ≥ 70 mL/min
* FEV_1 ≥ 60% by pulmonary function tests (PFTs)
* FVC ≥ 60% by PFTs
* DLCO ≥ 60% by PFTs
* For children who are unable to cooperate for PFTs all of the following criteria must be met:

  * No evidence of dyspnea at rest
  * No exercise intolerance
  * No requirement for supplemental oxygen therapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No HIV or uncontrolled fungal, bacterial, or viral infection

  * Fungal infection acquired during induction therapy allowed provided there is a significant response to antifungal therapy with minimal or no evidence of disease by CT scan
* Other concurrent immunosuppressants allowed
* No prior allogeneic or autologous stem cell transplantation
* No prior or concurrent voriconazole unless prior voriconazole therapy is completed or a different agent is substituted for voriconazole prior to study entry
* No concurrent grapefruit juice during sirolimus administration

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 146 (Actual)
Dates: Start 2007-03; Primary Completion 2011-05 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pulsipher, MD, Principal Investigator — Children's Oncology Group
Locations (50):
- United States (44):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - City of Hope Medical Center, Duarte, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Childrens Hospital of Orange County, Orange, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - University of California San Francisco Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Childrens Memorial Hospital, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kosair Children's Hospital, Louisville, Kentucky
  - Children's Hospital-Main Campus, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - New York Medical College, Valhalla, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (2):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (4):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec

REFERENCES:
- [Derived] Pulsipher MA, Carlson C, Langholz B, Wall DA, Schultz KR, Bunin N, Kirsch I, Gastier-Foster JM, Borowitz M, Desmarais C, Williamson D, Kalos M, Grupp SA. IgH-V(D)J NGS-MRD measurement pre- and early post-allotransplant defines very low- and very high-risk ALL patients. Blood. 2015 May 28;125(22):3501-8. doi: 10.1182/blood-2014-12-615757. Epub 2015 Apr 10. PMID 25862561
- [Derived] Pulsipher MA, Langholz B, Wall DA, Schultz KR, Bunin N, Carroll WL, Raetz E, Gardner S, Gastier-Foster JM, Howrie D, Goyal RK, Douglas JG, Borowitz M, Barnes Y, Teachey DT, Taylor C, Grupp SA. The addition of sirolimus to tacrolimus/methotrexate GVHD prophylaxis in children with ALL: a phase 3 Children's Oncology Group/Pediatric Blood and Marrow Transplant Consortium trial. Blood. 2014 Mar 27;123(13):2017-25. doi: 10.1182/blood-2013-10-534297. Epub 2014 Feb 4. PMID 24497539

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tacro-MTX/Sirolimus GVHD Prophylaxis Regimen | Tacro-MTX GVHD Prophylaxis
Started | 76 | 70
Completed | 64 | 66
Not Completed | 12 | 4
Not completed — Adverse Event | 3 | 0
Not completed — Physician Decision | 6 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — ineligible | 2 | 0
Not completed — Other | 0 | 2
Not completed — consent withdrawal | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacro-MTX/Sirolimus GVHD Prophylaxis Regimen | Tacro-MTX GVHD Prophylaxis | Total
Number analyzed (Participants) | 76 | 70 | 146
Age, Continuous [Median (Full Range); unit: Year] | 9 [1 to 20] | 10 [1 to 21] | 9 [1 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 59
  Male | 46 | 41 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 59 | 51 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 12 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 16 | 39
  Not Hispanic or Latino | 51 | 53 | 104
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 71 | 62 | 133
  Canada | 3 | 2 | 5
  Australia | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Estimated Percentage of Participants With Event Free Survival
Description: An event is defined as relapse or transplant-related mortality. Relapse is defined in section 3.3 study protocol.
Time Frame: at 2 years
Population: Two ineligible patients on experimental arm excluded from analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Experimental: Tacro-MTX/Sirolimus GVHD Prophylaxis
- Control: Tacro-MTX GVHD Prophylaxis
Arm/Group | Experimental | Control
Number analyzed (Participants) | 74 | 70
percentage of participants | 45 [34 to 60] | 54 [41 to 69]

2. Secondary Outcome: Rate of Relapses
Description: An event is defined as relapse.
Time Frame: At 2 years
Population: 2 ineligible patients on experimental arm excluded from analysis.Testing for recurrent malignancy in the blood, marrow or other sites will be used to assess relapse after transplantation. For the purpose of this study, relapse is defined by either morphological or cytogenetic evidence of ALL consistent with pre-transplant features.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 74 | 70
percentage of participants | 41 [29 to 57] | 33 [23 to 49]

3. Secondary Outcome: Estimated Transplant Related Mortality Percentage
Description: Death in a patient who had not relapsed after transplant is defined as transplant-related mortality event.
Time Frame: 100 days
Population: 2 ineligible patients on experimental arm excluded from analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 74 | 70
percentage of participants | 13 [7 to 24] | 6 [2 to 15]

4. Secondary Outcome: Estimated Rate of Acute Graft VS Host Disease (GVHD)
Description: Any grade acute graft vs host disease (defined in APPENDIX II study protocol).
Time Frame: At 200 days
Population: 2 ineligible patients on experimental arm excluded from analysis. Definition of Acute GVHD: APPENDIX II: COG STEM CELL COMMITTEE CONSENSUS GUIDELINES FOR ESTABLISHING ORGAN STAGE AND OVERALL GRADE OF ACUTE GRAFT VERSUS HOST DISEASE (GVHD) page 90-96 protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Experiemental: Tacro-MTX/Sirolimus GVHD Prophylaxis
Arm/Group | Experiemental | Control
Number analyzed (Participants) | 74 | 70
percentage of participants | 32 [22 to 45] | 49 [38 to 63]

5. Secondary Outcome: Estimated Rate of Overall Chronic Graft VS Host Disease
Description: Chronic graft vs host disease is defined in APPENDIX III of study protocol.
Time Frame: At 2 years
Population: 2 ineligible patients on experimental arm excluded from analysis. Definition of Chronic GVHD: APPENDIX III: DEFINING CHRONIC GRAFT VS. HOST DISEASE (FROM BMT CTN MOP SEPT. 2005) on page 97 protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 74 | 70
percentage of participants | 22 [14 to 36] | 27 [18 to 40]

6. Secondary Outcome: Relative Contribution of Resistance by Acute Lymphoblastic Leukemia (ALL) Blasts to Cytolytic Therapy (e.g., Chemotherapy/Irradiation) as a Cause of Relapse Post-transplantation
Description: An event is defined as relapse or transplant-related mortality.
Time Frame: Up to 1 year
Population: We made a large number of xenograft models but were not able to correlate resistance to rapamycin in mice with outcome on the trial with the numbers that we had. For this reason, no specific publications addressing this aim were put forward.
Arm/Group | Experiemental | Control
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Relative Contribution of ALL Blasts to the Donor Immune Response as a Cause of Relapse Post Transplantation (Correlating Development of aGVHD With Relapse)
Description: An event is defined as relapse; estimated probability of relapse.
Time Frame: At 1 year
Population: Number at risk among no aGVHD and number at risk among aGVHD at 1 year. The two treatment regimens were intended to be analyzed together (combined data), as pre-specified in the study protocol, therefore results are not reported for each Arm of study.
Measure: Number; unit: percentage of participants
Groups:
- All Patients: Relative contribution of ALL blasts to the donor immune response as a cause of relapse post transplantation (correlating development of aGVHD with relapse).
Arm/Group | All Patients
Number analyzed (Participants) | 67
percentage of participants
  Experienced aGVHD, later relapsed: number analyzed (Participants) | 35
  Experienced aGVHD, later relapsed | 5
  No aGVHD occurence, relapsed: number analyzed (Participants) | 32
  No aGVHD occurence, relapsed | 24

8. Secondary Outcome: Relative Contribution of ALL Blasts to the Donor Immune Response as a Cause of Relapse Pre-Transplantation (MRD)
Description: An event is defined as relapse; relapse risk is reported. Not able to be performed given the low numbers of blast samples available.
Time Frame: At 2 months
Population: The two treatment regimens were intended to be analyzed together (combined data), as pre-specified in the study protocol. However, we are not able to perform this analysis given the low numbers of blast samples available.
Groups:
- All Patients: Relative contribution of ALL blasts to the donor immune response as a cause of relapse pre transplantation (MRD)
Arm/Group | All Patients
Number analyzed (Participants) | 0

9. Secondary Outcome: Chimerism
Description: Evaluate the relative contribution of resistance by ALL blasts to the donor immune response as a cause of relapse post transplantation.
Time Frame: Up to 12 months
Population: We are not able to perform this analysis given the low numbers of blast samples available.
Arm/Group | Experiemental | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: SAE field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs / CAeRs). This study did not collect information about grade 1 and 2 AEs. The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs. 4 experimental patients were excluded (2 ineligible, 2 no data).
Arm/Group | Tacro-MTX/Sirolimus GVHD Prophylaxis Regimen | Tacro-MTX GVHD Prophylaxis
Serious Adverse Events (participants affected / at risk) | 9/72 | 5/70
Other Adverse Events (participants affected / at risk) | 38/72 | 30/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacro-MTX/Sirolimus GVHD Prophylaxis Regimen (N=72) | Tacro-MTX GVHD Prophylaxis (N=70)
Acute kidney injury (Renal and urinary disorders) | 1 | 2
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 1
Death NOS (General disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 2
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Multi-organ failure (General disorders) | 2 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
Vascular disorders - Other, specify (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacro-MTX/Sirolimus GVHD Prophylaxis Regimen (N=72) | Tacro-MTX GVHD Prophylaxis (N=70)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Anal pain (Gastrointestinal disorders) | 1 | 0
Anaphylaxis (Immune system disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 5 | 3
Ascites (Gastrointestinal disorders) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 2
Ataxia (Nervous system disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bladder infection (Infections and infestations) | 0 | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Capillary leak syndrome (Vascular disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Death NOS (General disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 2
Hypertension (Vascular disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 8 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Infections and infestations - Other, specify (Infections and infestations) | 6 | 1
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Localized edema (General disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 12 | 8
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 22 | 21
Pericardial effusion (Cardiac disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Platelet count decreased (Investigations) | 22 | 20
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
White blood cell decreased (Investigations) | 23 | 21

LIMITATIONS AND CAVEATS:
Outcome Measures 6, 7, 8 and 9 are exploring in nature and did not investigate the actual relapse rates of the 2 treatment regiments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval.